CLINICAL TRIAL: NCT03500185
Title: Effectiveness of Pelvic Floor Muscles Training in Group for Women With Urinary Incontinence: a Randomized Clinical Test
Brief Title: Effectiveness of Pelvic Floor Muscles Training in Group for Women With Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-0316
Record Dates: First submitted 2017-10-19; First posted 2018-04-18 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Urinary Incontinence
Keywords: Physiotherapy; Pelvic floor; Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PFMT in group (Experimental): Participants randomized to this group will perform the PFMT protocol in a group, with physiotherapeutic supervision, lasting 1 hour, in the Outpatient Clinic of Gynecology of Hospital of Clinics of Porto Alegre (HCPA), for a period of 3 months. You will also be instructed to perform exercises at home. After this period, they will be reassessed and will follow the same protocol for another 3 months now at home. After this period, they will be evaluated again.
  Interventions: Other: PFMT in group
- PFMT at home (Active Comparator): Randomized participants for this group will receive guidance on the home PFMT protocol on the day of the initial evaluation. They will be instructed to perform the exercises daily for a period of 3 months. After 3 months they will be re-evaluated and will follow the same protocol for another 3 months at home. After this period they will be evaluated again.
  Interventions: Other: PFMT at home

INTERVENTIONS:
Other: PFMT in group — Participants randomized to this group will perform the PFMT protocol in a group, with physiotherapeutic supervision, lasting 1 hour, in the Outpatient Clinic of Gynecology of Hospital of Clinics of Porto Alegre (HCPA), for a period of 3 months. You will also be instructed to perform exercises at home. After this period, they will be reassessed and will follow the same protocol for another 3 months now at home. After this period, they will be evaluated again.
  Arms: PFMT in group
Other: PFMT at home — Randomized participants for this group will receive guidance on the home PFMT protocol on the day of the initial evaluation. They will be instructed to perform the exercises daily for a period of 3 months. After 3 months they will be re-evaluated and will follow the same protocol for another 3 months at home. After this period they will be evaluated again.
  Arms: PFMT at home

SUMMARY:
The aim of the study is to compare the efficacy of a protocol, pelvic floor muscle training (PFMT), applied in a group and at home for urinary incontinence (UI) in women. Probably, the group-applied PFMT protocol is more effective in women with UI than the home protocol.

DETAILED DESCRIPTION:
Introduction: One of the female pelvic floor (PF) papers is to control urinary continence.

Changes in your PF function and structure can cause the dysfunction of the PF. Among these UI is more commonly reported and affects one-third of adult women and generates significant impact on the quality and life of these, including sexual activity. Among the possibilities to treat UI in a conservative manner, the PFMT should be recommended as an intervention of first-line treatment for women with such symptoms. Such training can be developed individually or in a group, just to be prescribed and performed 6-12 weeks to demonstrate such effectiveness. Nevertheless they are still scarce in the literature studies involving the PFMT, group and individual in application, that have validated and well-defined protocols and, in addition, protocols that are easy to understand and play by the patients.

Objective: The aim of the study is to compare the efficacy of a protocol of PFMT applied in a group and at home for UI in women.

Methodology: The study presents an experimental design type randomized blind clinical trial. The sample is not probabilistic for convenience, which shall contain the minimum number of 28 women in each group, obtained in the sample calculation. Women will be included from age 30 to 70 years who have had sexual intercourse in the last 12 months and who are able to understand the instruments, and sign the consent form. Women will be excluded with latex allergy, who have made treatment of pelvic radiotherapy, or are undergoing chemotherapy, women who had childbirth in the last 12 months which have participated in PFMT individually or in groups in the past six months. The assessment consists of a medical history form, which will include personal data; the evaluation of the function of PF is performed by the muscles pressure biofeedback apparatus which measures pressure peak contraction of the pelvic floor via a cuff connected to the pressure transducer; to assess the impact of UI on quality of life will use the International Consultation on Incontinence Questionnaire (ICIQ-SF); for evaluation of sexual function is used Pelvic Organ Prolapse Quiz / Urinary Incontinence Sexual Questionnaire (PISQ-12). Statistical analysis will be performed using the Shapiro-Wilk test to verify the normality of the data. Descriptive analysis of parametric data will be expressed as mean and standard deviation, and the nonparametric median and interquartile range. The qualitative variables are expressed as absolute and relative frequency. In the inferential analysis will be used for comparison of continuous variables parametric intragroup, ANOVA and non-parametric variables the Wilcoxon test. In the analysis of categorical variables will be used the McNemar test. As for the inferential analysis will be used for comparison of continuous variables parametric intergroup, ANOVA and non-parametric variables the Mann-Whitney test. In the analysis of categorical variables will be used chi-square test. For all analyzes will be of significance level of 5% (p ≤ 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Be female;
* Have urinary incontinence;
* Between 30 and 70 years old;
* Have had sexual intercourse in the last 6 months;
* Participants should understand the instruments used in the research;
* Accept to participate in the study and sign the Term of Free and Informed Consent.

Exclusion Criteria:

* Have allergy to latex;
* Have performed or are undergoing pelvic radiotherapy;
* Be performing chemotherapy treatment;
* Women who delivered during the last 12 months;
* Have participated in individual or group PFMT in the last 6 months;
* Have contraction of the pelvic floor muscles grade zero (0).

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Functionality of pelvic floor muscles | Evaluation after 24 weeks
  Capacity of voluntary contraction that reduces light and vaginal length, generating intravaginal pressure, in the case of this study evaluated by PERFECT Scale.

SECONDARY OUTCOMES:
Sexual function | Evaluation after 24 weeks
  A set of four successive stages: desire, arousal, orgasm and resolution, which have subjective, interpersonal, psychological, muscular and reflex characteristics, in the case of this study evaluated by the Pelvic Organ Prolapse / Urinary Incontinence Sexual Questionnaire (PISQ-12) .
Quality of life in urinary incontinence | Evaluation after 24 weeks
  The presence of urinary incontinence causes a substantial and substantial negative impact on the quality of life of women living with this symptom. This impact on quality of life can be measured by the International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF).

CONTACTS AND LOCATIONS:
Overall Officials: JOSÉ GERALDO LOPES RAMOS, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322